CLINICAL TRIAL: NCT05294809
Title: Effectiveness and Mechanisms of Change of Two Mobile Psychological Interventions in Reducing Depressive, Anxiety and Stress Symptoms: PsyPills and Online-Contingent Attention Training (OCAT)
Brief Title: Psychological Mobile Interventions to Reduce Distress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Babes-Bolyai University (Other)
Collaborators: Universidad Complutense de Madrid (Other)
Responsible Party: Principal Investigator, Sîrbu Vasile, PhD student, Babes-Bolyai University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 13.912 / 29.10.2021
Record Dates: First submitted 2022-02-23; First posted 2022-03-24 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Psychological Distress
Keywords: mobile mental health; mHealth; attention bias training; psychological distress; digital CBT; emotion regulation; functional reappraisal; rumination
MeSH Terms: conditions — Emotional Regulation; Rumination Syndrome

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of three conditions: 2 experimental conditions and an active control group.
Who Masked: Participant
Masking Description: Participants in all categories will be announced that they have received a mobile intervention aimed at distress reduction, without knowing the the rationale and specifics of each intervention. Outcomes will be assessed only by online questionnaires, so no assessor is involved.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- PsyPills (Experimental): The participants randomized in this condition will receive the mobile health application "PsyPills".
  Interventions: Behavioral: PsyPills
- OCAT (Experimental): The participants randomized in this condition will receive the mobile health application "OCAT".
  Interventions: Behavioral: Online-Contingent Attention Training, OCAT
- OCAT sham (Placebo Comparator): The active control group, which consists of the "fake" version of the OCAT intervention, by offering the same attentional training, without training and feedback on performance.
  Interventions: Behavioral: shamOCAT

INTERVENTIONS:
Behavioral: PsyPills — Prescribing personalized rational thinking strategies to change levels of dysfunctional emotionality.
  Arms: PsyPills
Behavioral: Online-Contingent Attention Training, OCAT — Facilitating the disengagement from negative content and engagement of positive one of personally relevant information by providing instruction and feedback on performance.
  Arms: OCAT
Behavioral: shamOCAT — The active control group, which consists of the "fake" version of the OCAT intervention, by offering the same attentional training, without training and feedback on performance.
  Arms: OCAT sham

SUMMARY:
Investigating the effectiveness of two mobile psychological interventions and the mechanisms of change involved in reducing the symptoms of depression, anxiety and stress, on an adult population with a mild to moderate level of symptoms (sub-clinical).

DETAILED DESCRIPTION:
The research design will be a 3-arm controlled clinical trial, with 4 waves of data collection. Once selected using a symptomatic screening questionnaire, participants will be randomly assigned to one of three conditions: 2 experimental conditions (PsyPills and OCAT) and an active control group (shamOCAT).

Measurements will be collected before allocation (baseline), during the intervention (through a momentary ecological assessment paradigm), at the end (post) and at an interval of one month after the intervention (follow-up). Among the constructs evaluated are symptomatic level, affectivity, cognitive processes, emotional regulation and attentional bias. All measurement steps will be collected online.

The interventions consist of an attentional training (Online-Contingent Attention Training, OCAT) which seeks to facilitate the disengagement from the negative content and the engagement on the positive of some personally relevant information by providing instructions and feedback on performance; and prescribing personalized rational thinking strategies to change the intensity of dysfunctional emotionality (PsyPills). The active control group consists of a "fake" version of OCAT (shamOCAT), by offering the same attentional training, without training and feedback on performance. All interventions are delivered in the form of smartphone applications.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old
* Have access and able to use a smartphone

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Actual)
Dates: Start 2022-06-12 (Actual); Primary Completion 2023-10-29 (Actual); Study Completion 2023-10-29 (Actual)

PRIMARY OUTCOMES:
Depressive, Anxiety, and Stress Symptoms | Baseline
  DASS-21, with scores from 0 to 63, higher scores meaning worse outcomes
Change from Baseline Depressive, Anxiety, and Stress Symptoms at 5 days | Mid of intervention (5 days)
  DASS-21, with scores from 0 to 63, higher scores meaning worse outcomes
Change from Baseline Depressive, Anxiety, and Stress Symptoms at 10 days | Post intervention (10 day)
  DASS-21, with scores from 0 to 63, higher scores meaning worse outcomes
Change from Baseline Depressive, Anxiety, and Stress Symptoms at 1 month | Follow-up (1 month)
  DASS-21, with scores from 0 to 63, higher scores meaning worse outcomes

SECONDARY OUTCOMES:
Functional Reappraisal | Baseline
  Acceptance, Putting into perspective and inversed scores of Catastrophizing subscales of CERQ-SF, with scores from 6 to 30, higher scores meaning better outcomes
Change from Baseline Functional Reappraisal at 5 days | Mid of intervention (5 days)
  Acceptance, Putting into perspective and inversed scores of Catastrophizing subscales of CERQ-SF, with scores from 6 to 30, higher scores meaning better outcomes
Change from Baseline Functional Reappraisal at 10 days | Post intervention (10 day)
  Acceptance, Putting into perspective and inversed scores of Catastrophizing subscales of CERQ-SF, with scores from 6 to 30, higher scores meaning better outcomes
Change from Baseline Functional Reappraisal at 1 month | Follow-up (1 month)
  Acceptance, Putting into perspective and inversed scores of Catastrophizing subscales of CERQ-SF, with scores from 6 to 30, higher scores meaning better outcomes
Positive Reappraisal | Baseline
  Positive reappraisal subscale of CERQ-SF, with scores from 2 to 10, higher scores meaning better outcomes
Change from Baseline Positive Reappraisal at 5 days | Mid of intervention (5 days)
  Positive reappraisal subscale of CERQ-SF, with scores from 2 to 10, higher scores meaning better outcomes
Change from Baseline Positive Reappraisal at 10 days | Post intervention (10 days)
  Positive reappraisal subscale of CERQ-SF, with scores from 2 to 10, higher scores meaning better outcomes
Change from Baseline Positive Reappraisal at 1 month | Follow-up (1 month)
  Positive reappraisal subscale of CERQ-SF, with scores from 2 to 10, higher scores meaning better outcomes
Rational and Irrational Beliefs | Baseline
  HABS-AV, with scores from 24 to 120, with higher scores meaning worse outcomes
Change from Baseline Rational and Irrational Beliefs at 5 days | Mid of intervention (5 days)
  HABS-AV, with scores from 24 to 120, with higher scores meaning worse outcomes
Change from Baseline Rational and Irrational Beliefs at 10 days | Post intervention (10 days)
  HABS-AV, with scores from 24 to 120, with higher scores meaning worse outcomes
Change from Baseline Rational and Irrational Beliefs at 1 month | Follow-up (1 month)
  HABS-AV, with scores from 24 to 120, with higher scores meaning worse outcomes
Rumination | Baseline
  Focus on thought/rumination subscale of CERQ-SF, with scores from 2 to 10, higher scores meaning worse outcomes
Change from Baseline Rumination at 5 days | Mid of intervention (5 days)
  Focus on thought/rumination subscale of CERQ-SF, with scores from 2 to 10, higher scores meaning worse outcomes
Change from Baseline Rumination at 10 days | Post intervention (10 days)
  Focus on thought/rumination subscale of CERQ-SF, with scores from 2 to 10, higher scores meaning worse outcomes
Change from Baseline Rumination at 1 month | Follow-up (1 month)
  Focus on thought/rumination subscale of CERQ-SF, with scores from 2 to 10, higher scores meaning worse outcomes
Functional and Dysfunctional Emotions | Baseline
  PAD, functional emotions subscale, with scores from 12 to 60, and dysfunctional emotions subscale, with scores from 14 to 70, with higher scores meaning worse outcomes
Change from Baseline Functional and Dysfunctional Emotions at 5 days | Mid of intervention (5 days)
  PAD, functional emotions subscale, with scores from 12 to 60, and dysfunctional emotions subscale, with scores from 14 to 70, with higher scores meaning worse outcomes
Change from Baseline Functional and Dysfunctional Emotions at 10 days | Post intervention (10 days)
  PAD, functional emotions subscale, with scores from 12 to 60, and dysfunctional emotions subscale, with scores from 14 to 70, with higher scores meaning worse outcomes
Change from Baseline Functional and Dysfunctional Emotions at 1 month | Follow-up (1 month)
  PAD, functional emotions subscale, with scores from 12 to 60, and dysfunctional emotions subscale, with scores from 14 to 70, with higher scores meaning worse outcomes
Attention bias | Baseline
  Engagement in positive information and inhibition of negative information web measures with an index of attention bias for processing positive vs. negative material computed by dividing the total fixation time on positive words by the total fixation time on emotional (positive and negative) words
Change from Baseline Attention Bias at 5 days | Mid of intervention (5 days)
  Engagement in positive information and inhibition of negative information web measures with an index of attention bias for processing positive vs. negative material computed by dividing the total fixation time on positive words by the total fixation time on emotional (positive and negative) words
Change from Baseline Attention Bias at 10 days | Post intervention (10 days)
  Engagement in positive information and inhibition of negative information web measures with an index of attention bias for processing positive vs. negative material computed by dividing the total fixation time on positive words by the total fixation time on emotional (positive and negative) words
Change from Baseline Attention Bias at 1 month | Follow-up (1 month)
  Engagement in positive information and inhibition of negative information web measures with an index of attention bias for processing positive vs. negative material computed by dividing the total fixation time on positive words by the total fixation time on emotional (positive and negative) words

OTHER OUTCOMES:
Experience Sampling Methods (ESM) questionnaire | During the intervention (3 times daily from day 1 to day 10)
  Items selected from the main scales, including 8 items for rational/irrational beliefs, 9 affective state items, 5 items from the subscales of interest of CERQ-SF, on a visual analog scale (VAS) format; the direction of scores is the same with those of the original scales and subscales from which th items are taken from

CONTACTS AND LOCATIONS:
Overall Officials: Oana David, Dr., Study Director — Babes-Bolyai University
Locations (1):
- Babes-Bolyai University, Cluj-Napoca, Romania